CLINICAL TRIAL: NCT06889649
Title: Prospective Study on the Efficacy and Safety of Stereotactic Ablative Body Radiotherapy Combined with Axitinib and Toripalimab in Recurrent or Metastatic Renal Cell Carcinoma
Brief Title: SABR Combined with Axitinib and Toripalimab in Recurrent or Metastatic RCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUFH-RCC-SABR-001
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Radiation Therapy; Targeted Therapy; Immunotherapy; Renal Cancer Metastatic
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy: SABR + Axitinib + Toripalimab (Experimental): Patients in this arm will receive a combination of Stereotactic Ablative Body Radiotherapy (SABR), Axitinib, and Toripalimab.
  SABR: Radiation dose of 6-10 Gy per fraction, administered in 5 fractions for peripheral lesions. For lesions near organs at risk, partial-SABR will be used. If neither SABR nor partial-SABR is feasible, moderate hypofractionated radiotherapy (MHFRT) with curative doses will be applied. Treatment duration is 1-5 weeks based on lesion location.
  Axitinib (oral, tablet): 5 mg twice daily for the study duration or until progression or intolerable side effects.
  Toripalimab (intravenous infusion): 240 mg every 3 weeks for the study duration or until progression or unacceptable toxicity.
  Treatment continues until disease progression, adverse events requiring discontinuation, or other study termination criteria are met
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy (SABR); Drug: TORIPALIMAB INJECTION(JS001 ); Drug: Axitinib (VEGF-TKI)

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiotherapy (SABR) — Radiation dose of 6-10 Gy per fraction, administered in 5 fractions for peripheral lesions. For lesions near organs at risk, partial-SABR will be used. If neither SABR nor partial-SABR is feasible, moderate hypofractionated radiotherapy (MHFRT) with curative doses will be applied.
Drug: TORIPALIMAB INJECTION(JS001 ) — Toripalimab (intravenous infusion):
  Dosage: 240 mg intravenously every 3 weeks. Frequency: Administered every 3 weeks for the duration of the study, until progression or unacceptable toxicity occurs or reach 2 years.
Drug: Axitinib (VEGF-TKI) — Axitinib (oral, tablet):
  Dosage: 5 mg orally twice daily. Frequency: Daily, for the duration of the study, with continuation during progression or until intolerable side effects occur.

SUMMARY:
This is a prospective, single-center clinical trial designed to evaluate the safety and efficacy of combining stereotactic ablative body radiotherapy (SABR) with the targeted therapy Axitinib and the immunotherapy Toripalimab in patients with recurrent metastatic renal cell carcinoma (RCC). Patients will receive a treatment regimen consisting of Axitinib, Toripalimab, and comprehensive multi-lesion SABR. The primary endpoint is Progression-Free Survival 1 (PFS1), and secondary endpoints include Progression-Free Survival 2 (PFS2), Overall Survival (OS), Local Control (LC), Objective Response Rate (ORR), and Disease Control Rate (DCR). Adverse events will be monitored according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0). The aim of this study is to explore a potentially more effective treatment combination for recurrent metastatic RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed renal cell carcinoma with recurrent metastatic lesions confirmed by PET/CT or other systemic imaging.
2. Patients with ≤5 metastatic lesions amenable to complete lesion coverage radiotherapy; or >5 lesions with at least 3 suitable for radiotherapy as evaluated by the radiotherapy and imaging departments.
3. Age between 18-80 years.
4. Expected survival of ≥12 weeks.
5. Measurable disease based on RECIST Version 1.1.
6. ECOG performance status of 0-2.

Exclusion Criteria:

1. History of anti-PD-1 or PD-L1 antibody therapy, or radiotherapy.
2. Use of corticosteroids or other immunosuppressants within 14 days before treatment.
3. Autoimmune diseases.
4. History of other malignancies.
5. History of surgery within 28 days before treatment.
6. Allergy to study drug components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival 1 (PFS1) | From the start of SABR treatment to the first disease progression, up to 2 years. This primary endpoint assesses how long patients survive without disease progression while receiving the combination therapy.
  PFS1 is defined as the time from the initiation of stereotactic ablative body radiotherapy (SABR) to the first occurrence of disease progression, as determined by radiological imaging (CT, MRI, or PET/CT) based on RECIST criteria. Disease progression is defined as an increase in the size of target lesions or the appearance of new lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the start of treatment to death or until the end of the study (up to 3 years). This secondary endpoint will help evaluate the overall survival benefits of the combined treatment over a longer period.
  Overall survival is defined as the time from the start of treatment (SABR combined with Axitinib and Toripalimab) to death from any cause.
Progression-Free Survival 2 (PFS2) | From the start of SABR treatment to the initiation of next-line treatment or death (an average of 3 year)
  PFS2 is defined as the time from the start of stereotactic ablative body radiotherapy (SABR) to the need for second-line treatment due to disease progression or clinical deterioration, or to death. This will be measured by assessing the time until the initiation of a next-line treatment regimen or the occurrence of death.

OTHER OUTCOMES:
Local Control (LC) | Through study completion, an average of 3 year
  Local Control is defined as the percentage of patients who have no evidence of disease progression in the irradiated lesions after treatment
Objective Response Rate (ORR) | From the start of treatment to the first radiological evaluation to the best response(an average of 6 months)
  Objective Response Rate is defined as the percentage of patients who achieve a complete response (CR) or partial response (PR)
Disease Control Rate (DCR) | From the start of treatment to the first disease progression, up to 2 years.
  Disease Control Rate is defined as the percentage of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu K, Ma MW, Gao XS, Li HZ, Chen JY, Li XY, Qin SB, Ren XY. Efficacy and safety of SABR/partial-SABR combined with axitinib and toripalimab in recurrent or metastatic renal cell carcinoma: Preliminary results from a prospective phase 2 trial. Oncol Lett. 2025 Jun 2;30(2):376. doi: 10.3892/ol.2025.15122. eCollection 2025 Aug. PMID 40503038